CLINICAL TRIAL: NCT00788567
Title: A Randomized, Open-label Study of the Achievement of a Mycophenolic Acid Therapeutic Window During Treatment With 2 Dosing Regimens of Oral CellCept Administered as a Component of Standard Immunosuppressive Therapy in Patients With Kidney Transplants
Brief Title: CLEAR Study - A Study of CellCept (Mycophenolate Mofetil) in Recipients of Kidney Transplants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18496
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: mycophenolate mofetil — 1
  Other Names: CellCept

SUMMARY:
This study will compare the efficacy and safety of 2 dosing regimens of oral CellCept administered as a component of standard immunosuppressive therapy in recipients of kidney transplants. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* recipients of a primary kidney transplant.

Exclusion Criteria:

* positive for HIV-1, human T-cell leukemia/lymphoma virus-1 (HTLV-1), or hepatitis B surface antigen;
* positive for hepatitis C virus, with moderate or severe liver disease;
* active malignancy or history of malignancy, excluding skin cancer (basal or squamous cell) that has been adequately treated;
* need for maintenance corticosteroids for another condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2005-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving therapeutic window by Day 5\n

SECONDARY OUTCOMES:
Efficacy: Achieving therapeutic window at Day 3, maintaining therapeutic window at day of discharge, Months 1, 3, and 6\nSafety: Renal function, opportunistic infections, malignancies, and adverse events\n

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (7):
- Canada (7):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Gourishankar S, Houde I, Keown PA, Landsberg D, Cardella CJ, Barama AA, Dandavino R, Shoker A, Pirc L, Wrobel MM, Kiberd BA. The CLEAR study: a 5-day, 3-g loading dose of mycophenolate mofetil versus standard 2-g dosing in renal transplantation. Clin J Am Soc Nephrol. 2010 Jul;5(7):1282-9. doi: 10.2215/CJN.09091209. Epub 2010 May 24. PMID 20498245